CLINICAL TRIAL: NCT02410369
Title: Phase II Study of S-588410 as Maintenance Monotherapy After Adjuvant Chemotherapy in Patients With Completely Resected Non-small- Cell Lung Cancer
Brief Title: Study of S-588410 After Adjuvant Chemotherapy for Completely Resected Non-small- Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo University (Other)
Collaborators: Kanagawa Cancer Center (Unknown); National Cancer Center Hospital East (Other); Shiga University of Medical Science (Unknown); Fukushima Medical University (Other); Hokkaido University (Other); Shionogi (Industry)
Responsible Party: Principal Investigator, Yataro Daigo, Project Professor, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMS2643; UMIN000016979 (Registry Identifier: UMIN)
Record Dates: First submitted 2015-03-04; First posted 2015-04-07 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Non-small- Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-588410 (Active Comparator): Subjects with HLA-A*2402 in the investigational arm will receive the subcutaneous administration of S-588410.
  Interventions: Drug: S-588410
- Placebo (Placebo Comparator): Subjects with HLA-A*2402 in the placebo arm will receive the subcutaneous administration of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-588410 — Following randomization, subjects with HLA-A*2402 in the investigational arm will receive the subcutaneous administration of S-588410.
  Arms: S-588410
Drug: Placebo — Following randomization, subjects with HLA-A*2402 in the investigational arm will receive the subcutaneous administration of Placebo.
  Arms: Placebo

SUMMARY:
In this clinical study, the investigators evaluate the efficacy and safety of S-588410 in patients who underwent an adjuvant chemotherapy after the complete resection of non-small-cell lung cancer.

DETAILED DESCRIPTION:
In this phase II trial, the investigators evaluate the efficacy and safety of S-588410 containing oncoantigens-derived HLA-A*2402-restricted epitope peptides in patients with HLA-A*2402 who underwent an adjuvant chemotherapy after the complete resection of non-small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received platinum-based adjuvant chemotherapy after the complete resection of lung cancer.
2. Pathologically determined non-small-cell lung cancer excepting the large cell neuroendocrine carcinoma and mixed type.
3. Patients with HLA-A*24:02.
4. Neither recurrence nor metastasis of non-small-cell lung cancer demonstrated by imaging tests within 6 weeks prior to the registration.
5. Possible to receive S-588410 within 12 weeks after the last adjuvant chemotherapy.
6. ECOG performance status 0 or 1 within 2 weeks prior to the registration.
7. Age over 20 years at time of consent acquisition.
8. The written informed consent provided by the patient.

Exclusion Criteria:

1. Other malignant diseases requiring treatment, excepting the cured cancer in-situ.
2. Concurrent treatment with anticancer drug, steroids, immunosuppressive agent, radiotherapy, immunotherapy, hyperthermia, or surgery.
3. Active and uncontrolled infectious disease.
4. Severe hepatic dysfunction, kidney dysfunction, cardiac disease, pulmonary disease, hematological disorder, or metabolic disease.
5. Coronary artery stenting within 6 months prior to registration.
6. Autoimmune disease.
7. HIV infection.
8. Registration within 4 weeks after the last adjuvant chemotherapy.
9. Laboratory values defined in the protocol within 2 weeks prior to registration.
10. Residual uncontrolled adverse events by adjuvant chemotherapy.
11. Eosinophilia within 28 days prior to registration. Past or active eosinophilic pneumonia or interstitial pneumonitis.
12. Past history of severe allergic reaction against drug, vaccine and biological agents.
13. Female patient in nursing or pregnancy.
14. Refusal of pregnancy conception.
15. Treated with the same peptide vaccines as S-588410.
16. Treated with another investigational drug within 28 days prior to registration or the period of 5 times of the drug half-life.
17. Decision of non-enrollment of the patients by principal investigator or physician-in-charge from the view point of patient's safety.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Relapse-free Survival Time as a Measure of Efficacy | 2 years

SECONDARY OUTCOMES:
Relapse-free Survival Rate after Randomization as a Measure of Efficacy | 1 and 2 years
Association between Relapse-free Survival Time and Induction of Cytotoxic T Lymphocytes Specific for Peptides | 2 years
Overall Survival Time as a Measure of Efficacy | 4 years
Overall Survival Rate after Randomization as a Measure of Efficacy | 1 and 2 years
Grade and Incidence of Adverse Events as a Measure of Safety and Tolerability | 4 years
Association between Overall Survival Time as a Measure of Efficacy and Gene Variation detected by Genomics Methods in Lymphocytes as a Predictive Biomarker | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Yataro Daigo, MD, PhD, Principal Investigator — Institute of Medical Science, The University of Tokyo
Locations (1):
- Institute of Medical Science, The University of Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harao M, Hirata S, Irie A, Senju S, Nakatsura T, Komori H, Ikuta Y, Yokomine K, Imai K, Inoue M, Harada K, Mori T, Tsunoda T, Nakatsuru S, Daigo Y, Nomori H, Nakamura Y, Baba H, Nishimura Y. HLA-A2-restricted CTL epitopes of a novel lung cancer-associated cancer testis antigen, cell division cycle associated 1, can induce tumor-reactive CTL. Int J Cancer. 2008 Dec 1;123(11):2616-25. doi: 10.1002/ijc.23823. PMID 18770861
- [Background] Hayama S, Daigo Y, Kato T, Ishikawa N, Yamabuki T, Miyamoto M, Ito T, Tsuchiya E, Kondo S, Nakamura Y. Activation of CDCA1-KNTC2, members of centromere protein complex, involved in pulmonary carcinogenesis. Cancer Res. 2006 Nov 1;66(21):10339-48. doi: 10.1158/0008-5472.CAN-06-2137. PMID 17079454
- [Background] Tomita Y, Yuno A, Tsukamoto H, Senju S, Kuroda Y, Hirayama M, Imamura Y, Yatsuda J, Sayem MA, Irie A, Hamada A, Jono H, Yoshida K, Tsunoda T, Daigo Y, Kohrogi H, Yoshitake Y, Nakamura Y, Shinohara M, Nishimura Y. Identification of immunogenic LY6K long peptide encompassing both CD4+ and CD8+ T-cell epitopes and eliciting CD4+ T-cell immunity in patients with malignant disease. Oncoimmunology. 2014 Mar 27;3:e28100. doi: 10.4161/onci.28100. eCollection 2014. PMID 25340007
- [Background] Kono K, Mizukami Y, Daigo Y, Takano A, Masuda K, Yoshida K, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Vaccination with multiple peptides derived from novel cancer-testis antigens can induce specific T-cell responses and clinical responses in advanced esophageal cancer. Cancer Sci. 2009 Aug;100(8):1502-9. doi: 10.1111/j.1349-7006.2009.01200.x. Epub 2009 May 14. PMID 19459850
- [Background] Mizukami Y, Kono K, Daigo Y, Takano A, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Detection of novel cancer-testis antigen-specific T-cell responses in TIL, regional lymph nodes, and PBL in patients with esophageal squamous cell carcinoma. Cancer Sci. 2008 Jul;99(7):1448-54. doi: 10.1111/j.1349-7006.2008.00844.x. Epub 2008 Apr 30. PMID 18452554
- [Background] Ishikawa N, Takano A, Yasui W, Inai K, Nishimura H, Ito H, Miyagi Y, Nakayama H, Fujita M, Hosokawa M, Tsuchiya E, Kohno N, Nakamura Y, Daigo Y. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res. 2007 Dec 15;67(24):11601-11. doi: 10.1158/0008-5472.CAN-07-3243. PMID 18089789
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873
- [Background] Daigo Y, Takano A, Teramoto K, Chung S, Nakamura Y. A systematic approach to the development of novel therapeutics for lung cancer using genomic analyses. Clin Pharmacol Ther. 2013 Aug;94(2):218-23. doi: 10.1038/clpt.2013.90. Epub 2013 May 8. PMID 23657161
- [Background] Daigo Y, Nakamura Y. From cancer genomics to thoracic oncology: discovery of new biomarkers and therapeutic targets for lung and esophageal carcinoma. Gen Thorac Cardiovasc Surg. 2008 Feb;56(2):43-53. doi: 10.1007/s11748-007-0211-x. Epub 2008 Feb 24. PMID 18297458